CLINICAL TRIAL: NCT05331378
Title: A Double-masked, Randomized, 2-armed Comparative Study of a Myopia Control Lens (Test Lens) Versus Single Vision Lens (Control Lens).
Brief Title: Clinical Evaluation of a Myopia Control Lens in Slowing Myopia Progression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WS10258
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-08

CONDITIONS: Myopia, Progressive; Myopia
Keywords: refractive error; eye disease; short-sightedness; children myopia; myopia progression
MeSH Terms: conditions — Myopia, Degenerative; Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, 2-armed, double-masked, monocenter, clinical trial, which consists of 6 visits across 1 year. The test myopia control lens will be compared with a single vision control lens in evaluating study objectives. After obtaining informed consent and assent, a comprehensive eye examination for screening will be done among approximately 80 myopic children between the age of 8-13 years old for eligibility. After randomization, the subjects will be back for dispensing of study spectacles and for baseline visit, where assessment of study spectacles, biometry, and instructions to use study spectacles were done. A follow up visit will be conducted in 3, 6 and 12 months time, in which the latter visit will also be the end of visit. All of which are non-contact and non-invasive to the eyes.
Who Masked: Participant, Investigator
Masking Description: Subjects (and their parents/guardians) will be masked to the lens assignment. Sibling of subjects must be excluded due to the noticeable differences between the test and control spectacle lenses Only the statistician will be unmasked when comparing the two lenses. The investigator who is responsible for randomization and allocation will also be unmasked. However, the primary outcome variables (spherical equivalent refraction & axial length) will be taken by masked investigators. To facilitate this, the subject will be led into the room(s) containing a biometer without their study spectacles by the unmasked investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test myopia control lenses (Experimental): A myopia control spectacle lenses (test lenses) will be given to 1 arm to wear for 12 months.
  Interventions: Device: Test myopia control lenses
- Single vision lenses (Other): A single vision spectacle lenses (control lenses) will be given to 1 arm to wear for 12 months.
  Interventions: Device: Single vision lenses

INTERVENTIONS:
Device: Test myopia control lenses — A myopia control spectacle lenses (test lenses) will be given to 1 arm to wear for 12 months.
  Arms: Test myopia control lenses
Device: Single vision lenses — A single vision spectacle lenses (control lenses) will be given to 1 arm to wear for 12 months.
  Arms: Single vision lenses

SUMMARY:
This is a monocenter, randomized, controlled, parallel-group, double-masked clinical trial to evaluate the effectiveness of test lens in slowing myopia progression with respect to axial length elongation at baseline compared to a single vision spectacle lens (control). A total of 80 children will be recruited where 40 subjects will be allocated either to wear test lenses (group 1) or control lenses (group 2) for 1 year through randomization.

DETAILED DESCRIPTION:
As myopia is a growing worldwide problem, it is important to better understand the range of possible treatments to slow the progression of myopia. Spectacle lenses with aspherical lenslets were shown to be effective in reducing myopia progression and axial length elongation in children in the previous clinical trial. A dose-dependent effect was demonstrated, with higher lenslet asphericity having greater myopia control efficacy.

This double masked parallel group study will test the safety and effectiveness of a test lens designed to modify the area and amount of myopic defocus on the retina without compromising vision. The study population includes children in Singapore aged 8 to 13 years (80 subjects) at the time of commencing treatment. As age of myopia onset is known to be an important factor in rate of myopia progression, subject age at the time of enrollment will be used to balance randomization. Axial length and spherical equivalent refraction will be the primary measure for myopia progression. Visual acuity will also be compared between test lenses and control lenses to determine the quality of vision using test lenses.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subject and guardian, fluent English spoken, willing to follow protocol and able to read, comprehend and sign the informed consent & assent form.
* Equal to or greater than 8 years and not older than 13 years at time of informed consent and assent.
* Spherical equivalent refractive error (SER) by manifest refraction between -0.75 and -4.75 D in each eye.
* Astigmatism, if present, of not more than 1.50 D.
* Difference in SER between the two eyes (Anisometropia) by manifest refraction not more than 1.00 D.
* Best corrected visual acuity in each eye equal to or better than +0.10 logMAR (≥ 20/25 as Snellen)
* Be in good general health based on his/her and parent's/guardian's knowledge. Absence of ocular disease with full ophthalmic examination. Without any ocular or systemic condition known to affect refractive status.
* History of myopia control intervention
* Absence of strabismus by cover test at near or distance wearing correction.
* Absence of amblyopia
* Without ocular or systemic medications which, in the investigator's opinion, may significantly affect pupil size, accommodation or refractive state.

Exclusion Criteria

* Vulnerability of subject
* Participation in any clinical study within 30 days of the Baseline visit.
* Sibling of existing participant of this study

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Axial Length | 12 months
  Change in ocular axial length (mm) measured using Lenstar Optical Biometer.

SECONDARY OUTCOMES:
Spherical Equivalent Refraction | 6 months and 12 months
  Change in spherical equivalent refraction (Dioptres) through manifest subjective refraction.
Axial Length | 6 months
  Change in ocular axial length (mm) measured using Lenstar Optical Biometer.
Carry-over Effect | 18 months and 24 months
  Change in ocular axial length (mm) measured using Lenstar Optical Biometer after switching to STELLEST™ lenses

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tan, Principal Investigator — Essilor R&D Centre Singapore
Locations (1):
- Essilor R&D Centre Singapore, Singapore, Singapore

REFERENCES:
- [Background] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039